CLINICAL TRIAL: NCT01615471
Title: Lose-Now-NC: Feasibility of a Large Group Format Community Weight Loss Program Coupled With Internet Support
Brief Title: Lose Now North Carolina Community Weight Loss Program
Acronym: Lose Now NC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Deborah F Tate, PhD, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LNNC2012
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Obesity
Keywords: Obesity; Lifestyle Intervention; Group treatment; Internet Intervention
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Large Group (Active Comparator): In person group sessions in large group format (up to 125 others)
  Interventions: Behavioral: Group weight loss with companion internet
- Small group (Active Comparator): Small group in person sessions (up to 25 other participants)
  Interventions: Behavioral: Group weight loss with companion internet

INTERVENTIONS:
Behavioral: Group weight loss with companion internet — Monthly in-person group sessions with an companion internet weight loss intervention

SUMMARY:
The Lose Now NC research study aims to determine feasibility by delivering a community based weight loss program for 4 months in Kannapolis, NC in a large group format compared with smaller group format, (recruiting approximately 225 participants from Mecklenburg and Cabarrus counties and randomizing them to large or small group in-person sessions coupled with an interim internet program) to examine reach and recruitment potential, pilot intervention procedures, collect process measures to determine satisfaction, adherence, attrition, and estimate weight loss for planning a larger trial.

DETAILED DESCRIPTION:
Cancer is the leading cause of death in North Carolina (NC); over 17,400 deaths were attributable to cancer in 2009. Obesity is also a widespread problem; 65% of NC adults were overweight or obese in 2009. Obesity has been linked to risk of several cancers, most notably breast and colon cancer, and also to decreased survival rates. Thus, due to the prevalence and linkage of obesity to major cancers, helping adults to lose weight is necessary to reduce cancer burden statewide.

Fortunately, modest weight losses of only 5 to 10 percent of total body weight have been shown to improve health and are achievable with behavioral lifestyle modification programs, considered the "gold standard" intervention. To date, weight loss via lifestyle modification has been shown to be more effective, and more cost-effective, than pharmaceutical intervention for reducing risk of chronic disease. However, these "gold standard" programs are very time and resource intensive; involving weekly face-to-face (F2F) sessions with groups of 10-20 participants for, at minimum, 16-24 weeks followed by bi-weekly contacts for up to 2 years. To combat this problem investigators, including those from this investigative team, have explored using the Internet to deliver weight loss programs. Internet programs are modestly effective producing 4-7% weight loss (at 6 months) or roughly ½ of what intensive F2F programs can achieve. Internet programs that involve substantial human contact via e-mail produce the best outcomes, yet limit dissemination, and those that involve only automated feedback suffer from low utilization over time. What may be optimal is a hybrid model involving fewer F2F visits coupled with an Internet program. We are currently investigating an alternative F2F approach whereby participants attend F2F visits once per month, as phase 1 of a 6-step, stepped care approach to treating obesity (R01 HL084400). The initial results are promising; at 3 months weight losses did not differ significantly between the monthly F2F approach and weekly F2F approach (-15.23 + 10.22 lbs. weekly vs. -12.32 + 10.26 lbs. monthly; p>.05). While the monthly program is ¼ of the visits of the standard treatment approach, the group size of 20 still severely limits dissemination. Delivering this monthly F2F approach in much larger groups (approximately 200 or more), coupled with an Internet program between sessions, may represent an effective and disseminable approach for achieving weight loss in NC communities.

A standard behavioral intervention based on the DPP and Premier trials will be adapted for this protocol. Behavioral weight control approaches are founded on teaching skills and providing the support necessary to enable participants to adopt lower calorie diets (e.g., 1500-2000 kcals per day based on starting weight) and moderate physical activity (e.g., walking) to produce energy deficits necessary to produce modest weight losses of 1-2 lbs per week. Based on findings from the focus groups and review of study design and expectations from the funding source to conduct pilot research that will lead to future funding and publishable findings, the main intervention has been finalized (since initial IRB submission). The intervention will consist of randomization to either Large Group + Internet or Small Group + Internet interventions. The main difference between the two study groups will be the size of the monthly group sessions. The internet program delivered in between monthly group sessions will be identical. Group sessions will occur at the Nutrition Research Institute (NRI) on a monthly basis in months 1 - 4. The internet program will be used between group sessions. The monthly sessions will begin with an individual, private, weigh-in, followed by a group session. One treatment arm will have large group sessions with interactive features and audience participation. The large groups will be comprised of approx. 125 participants, last approximately 1 hour, and be facilitated by a weight loss expert (dietitian, psychologist, exercise physiologist). The other treatment arm will have small group sessions and will consist of approx. 25 participants and will follow traditional behavioral weight control group session protocol with facilitation by the above named-experts. Participants will be encouraged to enroll in the study with up to two friend or family member support partners who are also meet eligibility criteria. Support partners will be randomized to the same treatment arm. The F2F sessions are coupled with a comprehensive Internet program tested previously by Tate et al that provides the self-monitoring tools, tailored automated behavioral feedback, tailored lifestyle content (lessons) resources, and social support (e.g. online message board) that participants will be encouraged to use in between monthly sessions.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age. Older adults have more medical co-morbidities; since this community program has minimal face-to-face supervision, individuals age >65 will be ineligible.
2. Body mass index (BMI) greater than 25.0 kg/m2.
3. Access to the internet on at least a weekly basis.
4. Ability to read, write and speak English.
5. Ability to attend 4 monthly group sessions and 2 assessment visits (baseline and follow-up) at the Nutrition Research Institute.
6. Possession and usage of an internet e-mail address or willingness to sign up for a free email account (e.g., gmail)

Exclusion Criteria:

1. Pregnancy during the previous 3 months, or planned pregnancy in the folliowing 6 month (study period including assessments and treatment).
2. Current participation in another weight loss study or program (including weight loss medication) and unwilling to discontinue participation for the duration of the study.
3. Insulin treatment for diabetes mellitus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Weight change | 4 months
  Change in weight from baseline to 4 months

SECONDARY OUTCOMES:
Diet | 4 months
  Change in diet as assessed by ASA 24
Physical Activity | 4 months
  Change in Physical Activity as assessed by Paffenbarger Exercise Questionnaire
Lipids | 4 months
  Change in lipids
Hemoglobin A1c | 4 months
  Change in HbA1c
Blood Pressure | Baseline to 4 months
  Change in Blood Pressure from Baseline to 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Tate DF, Valle CG, Crane MM, Nezami BT, Samuel-Hodge CD, Hatley KE, Diamond M, Polzien K. Randomized trial comparing group size of periodic in-person sessions in a remotely delivered weight loss intervention. Int J Behav Nutr Phys Act. 2017 Oct 23;14(1):144. doi: 10.1186/s12966-017-0599-3. PMID 29061153